CLINICAL TRIAL: NCT00252759
Title: A Nested Case-control Study to Determine the Relative Risk of and Risk Factors for Interstitial Lung Disease in a Cohort of NSCLC Patients Treated With and Without Gefitinib
Brief Title: Iressa Case Control Study in Japan
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: D791AL00002; V-15-33; OZV1533
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purposes of this study are:

* To estimate the relative risk of ILD in advanced/recurrence NSCLC patients treated with gefitinib as compared to other chemotherapy treatment, and to assess the risk factors for ILD in advanced/recurrence NSCLC patients undergoing treatment
* To provide an estimate of the incidence of ILD in a group of advanced/recurrence NSCLC patients undergoing treatment

ELIGIBILITY:
Inclusion Criteria:

* Advanced/recurrence NSCLC patients who have had one or more chemotherapy regimens.
* Patients who are to be treated with gefitinib or chemotherapy
* Cohort: All advanced/recurrence NSCLC patients participating in this post-marketing clinical study

Exclusion Criteria:

* Patients judged by the investigator(s) to have ILD (provisional cases) among those registered in the cohort OR Randomly selected patients without ILD (controls) for each provisional case
* Case-control study: Patients enrolled in the case-control study; all consenting patients with ILD as cases and approximately 4 times as many consenting patients without ILD as controls randomly selected from the cohort

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2003-11; Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Japan Medical Director, MD, Study Director — AstraZeneca
Locations (44):
- Japan (44):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Okazaki, Aichi-ken
  - Research Site, Toyoake, Aichi-ken
  - Research Site, Imba-gun, Chiba
  - Research Site, Kashiwa, Chiba
  - Research Site, Matsuyama, Ehime
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kitakyushu, Fukuoka
  - Research Site, Gifu, Gifu
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Asahikawa, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Akashi, Hyōgo
  - Research Site, Kobe, Hyōgo
  - Research Site, Kanazawa, Ishikawa-ken
  - Research Site, Isehara, Kanagawa
  - Research Site, Sagamihara, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Kyoto, Kyoto
  - Research Site, Sendai, Miyagi
  - Research Site, Nagasaki, Nagasaki
  - Research Site, Ōmura, Nagasaki
  - Research Site, Tenri, Nara
  - Research Site, Niigata, Niigata
  - Research Site, Okayama, Okayama-ken
  - Research Site, Ginowan, Okinawa
  - Research Site, Habikino, Osaka
  - Research Site, Izumisano, Osaka
  - Research Site, Osaka, Osaka
  - Research Site, Sakai, Osaka
  - Research Site, Sayama, Osaka
  - Research Site, Toyonaka, Osaka
  - Research Site, Tokyo, Ota
  - Research Site, Ōtsu, Shiga
  - Research Site, Sunto-gun, Shizuoka
  - Research Site, Bunkyo-ku, Tokyo
  - Research Site, Bunkyo, Tokyo
  - Research Site, Kiyose, Tokyo
  - Research Site, Minato-ku, Tokyo
  - Research Site, Mitaka, Tokyo
  - Research Site, Shinjuku, Tokyo
  - Research Site, Toshima-ku, Tokyo
  - Research Site, Toyama, Toyama

REFERENCES:
- [Derived] Kawata T, Higashimori M, Itoh Y, Tomkinson H, Johnson MG, Tang W, Nyberg F, Jiang H, Tanigawara Y. Gefitinib exposure and occurrence of interstitial lung disease in Japanese patients with non-small-cell lung cancer. Cancer Chemother Pharmacol. 2019 May;83(5):849-858. doi: 10.1007/s00280-019-03788-4. Epub 2019 Feb 14. PMID 30762084